CLINICAL TRIAL: NCT07236866
Title: Prospective, Single-center Interventional Study to Assess the Reliability of the GRAMPA Score, Measuring the Graduation of Motor Abilities of the Elderly Patients Hospitalised
Brief Title: Evaluation of GRAMPA Score Measuring Motor Abilities of Elderly Patients
Acronym: GRAMPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Mutualiste de Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GRAMPA; Numero RCB (Other: 2025-A00650-49)
Record Dates: First submitted 2025-06-27; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Geriatric Assessment
Keywords: motor skills; rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scales Motricity (Experimental): The motor skills will be assessed using the GRAMPA scale and compared with the scales usually used in current practice: the minimum motor test (TMM) and the Katz scale (ADL).
  The GRAMPA scale will be carried out :
  * At admission
  * During the hospitalisation by two different physiotherapist
  * At discharge
  Interventions: Other: GRAMPA scale

INTERVENTIONS:
Other: GRAMPA scale — The GRAMPA scale will be carried out for every patient.
  The patient will be asked to do the following basic movement, in an order defined by the physiotherapist:
  * Get back into bed
  * Turn on the side in bed
  * Sit on the edge of the bed
  * Stand up
  * Move around the room
  * Sitting up
  * Getting back into bed
  It takes around 5 to 10 minutes to complete the scale

SUMMARY:
In the field of geriatrics, the Standardized Geriatric Approach (SGA) which is the benchmark for assessing elderly patients, consists of evaluating the medical, psychological and functional capacity dimensions of the elderly subject, among others.

After a review of the literature, investigators were unable to find any scales that could study the ability to perform basic movements in a comprehensive and graded manner.

Scores that do assess certain aspects of motor abilities are not comprehensive, and are often based on self-reporting by the elderly or their relatives :

* The AGGIR grid assesses dependency on the basis of activities performed or not performed. In addition, all basic movements are grouped together in a single item, which does not provide detailed information on the capabilities of elderly people.
* The ADL score assesses activities of daily living, based on what patients declare. Only one item concerns basic movements, without detailing them.
* The Tinetti score and Time up and go do not assess all basic movements, and require the patient to be able to stand to provide relevant information, whereas many geriatrics patients are unable to stand.

Thus, investigators created a score to assess motor abilities more comprehensively that will include the following basic movements:

* Getting up in bed
* Turning on one side in bed
* Sitting at the edge of the bed
* Stand up
* Move around a small perimeter (bedroom)
* Sitting up
* Return to bed

The main objective is to evaluate of this study is to determine the inter-rater reliability of the GRAMPA score in elderly patients hospitalized in a geriatric rehabilitation department.

DETAILED DESCRIPTION:
In the field of geriatrics, the Standardized Geriatric Approach (SGA) which is the benchmark for assessing elderly patients, consists of evaluating the medical, psychological and functional capacity dimensions of the elderly subject, among others. This approach is defined as a "multidimensional and interdisciplinary diagnostic process that seeks to assess the medical, psychological and functional capacity of the frail elderly person, with the aim of developing a coordinated and integrated long-term treatment and follow-up plan".

Mobility or functional capacity, an essential component of AGS, is generally studied in terms of balance, walking and basic movement, as in the Tinetti tests, the Timed up and go or walking speed. According to the French National Authority for Health (HAS), "the ability to perform basic movements largely determines the level of physical dependence. The important stages in assessing mobility and the quality of the strategies used are: raising in bed, turning on one side in bed, getting out of bed, moving from sitting to standing and from standing to sitting'.

After a review of the literature, investigators were unable to find any scales that could study the ability to perform basic movements in a comprehensive and graded manner. The Minimum Motor Test (MMT), a score created in 2005 with the aim of observing motor abilities and establishing rehabilitation objectives for patients suffering from psychomotor maladjustment syndrome, does not allow exhaustive evaluation of basic movements and is not very sensitive for distinguishing between two patients unable to hold the standing position (15 items /20 requiring standing). In particular, it does not include bed raising and sit-to-stand transfers. The test is based on clinical observations using two scoring levels: if the answer to the question asked is 'yes', the score awarded is 1; if the answer is 'no', the score awarded is 0. The maximum total score that can be obtained is 20. A high score means that good physical ability has been retained.

The AGGIR grid assesses dependency on the basis of activities performed or not performed. In addition, all basic movements are grouped together in a single item, which does not provide detailed information on the capabilities of elderly people.

The Activities of Daily Living (ADL) assesses independence in activities of daily living in the broadest sense, but does not specifically target functional motor skills. A score of 6 determines the maximum level of autonomy. The overall score varies from 0 (totally dependent) to 6 (best possible independence). Measuring ADLs is relevant for all elderly people, regardless of where they live.

Thus, investigators created a score, the GRAMPA score, to assess motor abilities more comprehensively that will include the following basic movements:

* Getting up in bed
* Turning on one side in bed
* Sitting at the edge of the bed
* Stand up
* Move around a small perimeter (bedroom)
* Sitting up
* Return to bed

In the GRAMPA score, these basic movements are characterised according to 3 grades of autonomy:

* Unassisted: The patient carries out the basic movement alone, without technical aid or verbal guidance.
* Partial assistance: The patient needs technical assistance, i.e. equipment, and/or verbal guidance to carry out the basic movement.
* Significant assistance: The patient needs human assistance to carry out the basic movement, i.e. as soon as the carer puts his/her hands on the patient to mobilise or support him/her, and/or the carer handles the heavy equipment needed to carry out the transfer.

Investigators believe that the GRAMPA score (GRaduation de l'Autonomie Motrice des Personnes Agées) would be a better reflection of the motor abilities of elderly subjects, by studying their ability to move in a restricted environment (e.g. a hospital room).

A more accurate estimate of basic functional motor skills would help to improve communication between healthcare professionals and optimise treatment by adapting strategies to the patient's level of functional autonomy (patient dependence in terms of equipment layout, rehabilitation objectives and limiting iatrogenic dependence).

As the metrological qualities of the score have not been validated, it will not be used to modify the management of patients included in the study.

There will therefore be no significant benefit or risk for participating patients.

Patients' motor skills are information that is communicated very regularly between healthcare professionals, and which is essential for helping patients regain their independence and organising care in a rehabilitation department. In particular, this information can be used to choose the technical aids best suited to patients' autonomy, or to decide on the possibility of a return home.

In particular, this score would enable better inter-professional communication about patients' functional abilities, leading to improved conditions for patient care by professionals.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 75 years
2. Patients hospitalised in the medical care and rehabilitation department of the Groupe Hospitalier Mutualiste de Grenoble.
3. Comprehension of the French language (understanding of instructions)
4. Signature of free and informed consent

Exclusion Criteria:

1. Patients whose sensory and/or mental capacities do not allow them to understand the instructions for carrying out transfers.
2. Patients with medical or surgical contraindications making it impossible to carry out transfers.
3. Patients under legal protection or unable to express their consent.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Assess the inter-rater reliability of the Motor Autonomy Assessment for the Elderly (GRAMPA) score. | Peri-interventional
  Intra-class correlation coefficient (ICC). The score will therefore be calculated by 2 different professionals on the same patient during hospitalisation.
  Score total GRAMPA [0;14] , Score =0 significant help, Score [1-7] = partial assistance, Score [8-14] = unaided

SECONDARY OUTCOMES:
Assess the convergent validity of the GRAMPA score against two established scales: Mini Moteur Test and Activities of Daily Living. | Baseline
  Correlation coefficient calculated between the GRAMPA score and each of the two scales Total TMM score [0;20] A high score means good physical; ADL Score 6=independent, 4=moderate impairment, 0= very dependent
Assess the convergent validity of the GRAMPA score against two established scales: Mini Moteur Test and Activities of Daily Living. | the end of the study i.e. 3 weeks on average
  Correlation coefficient calculated between the GRAMPA score and each of the two scales Total TMM score [0;20] A high score means good physical; ADL Score 6=independent, 4=moderate impairment, 0= very dependent

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble, Isere
  - Groupe Hospitalier Mutualiste, Grenoble, Isere

IPD SHARING:
Plan to Share IPD: No